CLINICAL TRIAL: NCT06674382
Title: Haploidentical Hematopoietic Stem Cell Transplantation for the Treatment of Myelofibrosis: A Prospective, Single-center Study
Brief Title: Haplo-HSCT for Myelofibrosis
Acronym: HHM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Yuqian, Associate Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB400-001; Peking University (Registry Identifier: Peking University)
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Myelofibrosis
Keywords: Haplo-HSCT; myelofibrosis; MF
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Haplo-SCT group (Experimental): Patients in this group will undergo haploidentical hematopoietic stem cell transplantation for the treatment of myelofibrosis.
  Interventions: Procedure: Haploidentical hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Haploidentical hematopoietic stem cell transplantation — This is a single-arm study in which all patients will undergo haploidentical hematopoietic stem cell transplantation for the treatment of myelofibrosis.
  Pre-transplant Evaluation:
  Evaluation includes status of primary Disease, donor specific antibodies (DSA), organ function (assessments for heart, liver, lungs, kidneys, and the nervous system), and Spleen size.
  Transplantation Protocol:
  Conditioning Regimen:
  Dac/TT/Bu/Flu/ATG regimen:
  Decitabine 100 mg/m², on day -12. Thiotepa (TT) 5 mg/kg/day, on days -11 and -10. Busulfan 0.8 mg/kg body weight, every 6 hours, on days -8 to -6. Fludarabine 30 mg/m², once daily, on days -6 to -2. Anti-thymocyte globulin (ATG) 2.5 mg/kg body weight, once daily, on days -5 to -2.
  Transplant Donor: Haploidentical donor. GVHD (Graft-versus-Host Disease) Prophylaxis Regimen: Cyclosporine, mycophenolate mofetil, and short-course methotrexate for GVHD prevention.
  Graft:
  Target MNC (Mononuclear Cells): 6-8 × 10⁸/kg. Target CD34+ stem cells: 5 × 10⁶/kg

SUMMARY:
Myelofibrosis (MF) is a myeloproliferative neoplasm causing bone marrow failure and high risk of leukemia transformation. JAK2 inhibitors improve symptoms but do not cure MF. Allogeneic stem cell transplantation (allo-HSCT) is the only potential cure, though limited donor availability restricts access. Haploidentical transplantation shows promise but associated with higher graft failure and treatment related mortality. We recently developed a novel regimen of haplo-SCT for MF. This study aims to investigate this novel protocol in a prospective trial to improve MF outcomes.

DETAILED DESCRIPTION:
Myelofibrosis (MF) is a myeloproliferative neoplasm characterized by clonal proliferation of hematopoietic stem cells, reactive hyperplasia of bone marrow stromal cells, and secondary inflammation and fibrosis, leading to progressive bone marrow failure and a high risk of acute myeloid leukemia transformation, with a median survival of about 6 years. While JAK2 inhibitors like ruxolitinib have been approved to improve symptoms and survival in MF patients, they do not provide a cure. Allogeneic stem cell transplantation (allo-HSCT) remains the only potential cure, but limited availability of matched sibling and unrelated donors often prevents patients from receiving this treatment. Haploidentical stem cell transplantation has shown good efficacy in leukemia but is less studied in MF, possibly due to concerns about graft failure, complications, and high transplant-related mortality. Our team has applied a novel haploidentical transplantation protocol for treating MF, which has shown promising results in preliminary observations. This study aims to further validate the effectiveness of this protocol through a prospective clinical trial, potentially establishing an effective approach for HSCT in MF and improving overall transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primary disease type: Myelofibrosis (including primary myelofibrosis and myelofibrosis secondary to polycythemia vera or essential thrombocythemia).
* No matched sibling donor or unrelated donor, with the availability of a haploidentical donor.
* Signed informed consent.

Exclusion Criteria:

1. Active infection
2. Very poor performance status (ECOG score > 2)
3. Estimated survival time < 30 days
4. Patient or family unable to cooperate
5. Considered unsuitable after discussion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of Good graft function at day 60 | Assessment at 60 days post-transplantation
  The cumulative incidence of achieving both neutrophil engraftment and platelet engraftment at day 60 after Hematopoietic stem cell transplantation, independent of transfusion and granulocyte growth factor support, using competing risk model.

SECONDARY OUTCOMES:
Transplant-related mortality | From baseline assessment at enrollment to the follow-up assessment at 36 months post-treatment.
  TRM is defined as death due to any transplantation-related cause other than disease relapse. Transplant-related mortality will be calculated using a competing risks model.
overall survival | From baseline assessment at enrollment to the follow-up assessment at 36 months post-treatment.
  The time from hematopoietic stem cell transplantation to death from any cause in patients with myelofibrosis. Overall survival will be calculated using the Kaplan-Meier method.
Cumulative Incidence of Relapse | From baseline assessment at enrollment to the follow-up assessment at 36 months post-treatment.
  Relapse was defined as disease recurrence. The criteria for relapse include:
  1. Increase in age-adjusted cellularity and abnormal M: E ratio.
  2. Megakaryocytic abnormalities typical of MF (pleomorphism, hyperchromatic, cloud-like nuclei and megakaryocytic clusters).
  3. Increase in grade of reticulin/collagen fibrosis (it should be borne in mind that the previously formed new bone usually takes a long time to be resorbed/resolved and that this should not therefore be used in grading post-transplant unless its density is significantly greater than the pre-transplant biopsy or there is active evidence of continuing new bone deposition).
Incidence of GVHD | From baseline assessment at enrollment to the follow-up assessment at 36 months post-treatment.
  The incidence refers to the rate at which new cases of GVHD occur within a timeframe. Acute GVHD was classified as symptom presentation before 100 days after alloHCT and chronic GVHD was classified as symptom presentation >100 days after alloHCT. Each organ (skin, liver, and gut) was staged 1 through 4 for Acute (a) GVHD according to modified criteria based on the schema of the Mount Sinai Acute GVHD International Consortium (MAGIC), and patients were also assigned a grade of acute GVHD (I through IV) based on overall severity. Chronic (c) GVHD was graded in accordance with the National Institutes of Health (NIH) Chronic Graft-versus-Host Disease Consensus Criteria.
Disease-free survival | From baseline assessment at enrollment to the follow-up assessment at 36 months post-treatment.
  The time from hematopoietic stem cell transplantation to the first occurrence of disease relapse, progression, or death from any cause in patients with myelofibrosis.
Neutrophil Engraftment | From baseline assessment at enrollment to the follow-up assessment at 60 days post-treatment.
  The time to neutrophil engraftment was defined as the first of three consecutive days with an ANC > 0.5 × 109/L.
Platelet Engraftment | From baseline assessment at enrollment to the follow-up assessment at 60 days post-treatment.
  The time to platelet engraftment was defined as the first of seven consecutive days with a platelet count >20 × 109/L without transfusion support.
Graft failure | From baseline assessment at enrollment to the follow-up assessment at 28 days post-treatment.
  Primary GF is defined by an ANC<0.5×109/l by day +28 following stem cell infusion, Hb <80 g/L and platelets <20×109 /L.Secondary GF is currently deﬁned by EBMT criteria as the presence of an ANC<0.5×109/L occurring after initial engraftment and not related to relapse, infection or drug toxicity.
Toxicity of conditioning | From baseline assessment at enrollment to the follow-up assessment at 30 days post-treatment.
  Toxicity of conditioning within 30 days of Hematopoietic Stem Cell Transplantation (HSCT) can be graded according to Common Terminology Criteria for Adverse Events (CTCAE):
  1. Grade 1: Mild toxicity that does not require medical intervention.
  2. Grade 2: Moderate toxicity that may require medical intervention.
  3. Grade 3: Severe toxicity that requires significant medical intervention, hospitalization, or results in lasting effects.
  4. Grade 4: Life-threatening toxicity, potentially requiring intensive care.
  5. Grade 5: Death caused by the toxicity reaction.
Grade of Bone Fibrosis | From baseline assessment at enrollment to the follow-up assessment at 12 months post-treatment.
  The degree of bone marrow fibrosis as assessed by histopathological examination, categorized according to The European Consensus on grading of bone marrow fibrosis in patients with myelofibrosis after hematopoietic stem cell transplantation.
Spleen Response | From baseline assessment at enrollment to the follow-up assessment at 12 months post-treatment.
  The change in spleen size, typically measured by imaging (e.g., ultrasound, CT scan), after hematopoietic stem cell transplantation, categorized as complete response, partial response, or no response according to the response criteria of IWG-MRT and ELN:
  * Complete Response (CR): The spleen is no longer palpable or measurable by imaging after treatment, indicating a full resolution of splenomegaly.
  * Partial Response (PR): A significant reduction in spleen size, typically defined as a reduction of at least 35% in spleen volume or a decrease in palpable spleen size.
  * No Response (NR): No reduction in spleen size, or the spleen size remains stable or worsens.
  * Progressive Disease (PD): The spleen increases in size after treatment, indicating worsening of splenomegaly.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Polverelli N, Hernandez-Boluda JC, Czerw T, Barbui T, D'Adda M, Deeg HJ, Ditschkowski M, Harrison C, Kroger NM, Mesa R, Passamonti F, Palandri F, Pemmaraju N, Popat U, Rondelli D, Vannucchi AM, Verstovsek S, Robin M, Colecchia A, Grazioli L, Damiani E, Russo D, Brady J, Patch D, Blamek S, Damaj GL, Hayden P, McLornan DP, Yakoub-Agha I. Splenomegaly in patients with primary or secondary myelofibrosis who are candidates for allogeneic hematopoietic cell transplantation: a Position Paper on behalf of the Chronic Malignancies Working Party of the EBMT. Lancet Haematol. 2023 Jan;10(1):e59-e70. doi: 10.1016/S2352-3026(22)00330-1. Epub 2022 Dec 6. PMID 36493799
- [Result] Cervantes F, Dupriez B, Passamonti F, Vannucchi AM, Morra E, Reilly JT, Demory JL, Rumi E, Guglielmelli P, Roncoroni E, Tefferi A, Pereira A. Improving survival trends in primary myelofibrosis: an international study. J Clin Oncol. 2012 Aug 20;30(24):2981-7. doi: 10.1200/JCO.2012.42.0240. Epub 2012 Jul 23. PMID 22826273
- [Result] Gangat N, Tefferi A. Myelofibrosis biology and contemporary management. Br J Haematol. 2020 Oct;191(2):152-170. doi: 10.1111/bjh.16576. Epub 2020 Mar 20. PMID 32196650